CLINICAL TRIAL: NCT00957112
Title: The Efficacy of Acupuncture and Self-acupuncture in Managing Cancer-related Fatigue in Breast Cancer Patients: a Pragmatic Randomised Trial
Brief Title: Acupuncture or Self-Acupuncture in Managing Cancer-Related Fatigue in Women Who Have Received Chemotherapy for Stage I, Stage II, or Stage IIIA Breast Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Manchester (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Supportive Care
Other Study IDs: CDR0000649750; UM-ASA; EU-20970
Record Dates: First submitted 2009-08-11; First posted 2009-08-12 (Estimated); Last update posted 2013-08-26 (Estimated); Status verified 2009-08

CONDITIONS: Anxiety Disorder; Breast Cancer; Depression; Fatigue
Keywords: anxiety disorder; depression; fatigue; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer
MeSH Terms: conditions — Anxiety Disorders; Breast Neoplasms; Depression; Fatigue | interventions — Acupuncture Therapy

ARMS (5):
- Arm I (Experimental): Patients undergo a 20-minute acupuncture session once a week for 6 weeks. Patients also receive written information about fatigue and its possible management.
  Interventions: Procedure: acupuncture therapy
- Arm II (No Intervention): Patients receive standard care. They also receive written information about fatigue as in arm I.
  Interventions: Procedure: standard follow-up care
- Arm A (Experimental): Patients receive treatment as in arm I for 4 more weeks.
  Interventions: Procedure: acupuncture therapy
- Arm B (No Intervention): Patients receive standard care as in arm II for 4 more weeks.
  Interventions: Procedure: standard follow-up care
- Arm C (Experimental): Patients learn to self-acupuncture and do so weekly for 4 more weeks.
  Interventions: Procedure: acupuncture therapy

INTERVENTIONS:
Procedure: acupuncture therapy — Patients undergo therapist-acupuncture with or without self-acupuncture
  Arms: Arm A; Arm C; Arm I
Procedure: standard follow-up care — Patients receive standard care
  Arms: Arm B; Arm II

SUMMARY:
RATIONALE: Acupuncture may help relieve fatigue caused by breast cancer. It is not yet known whether acupuncture is more effective than self-acupuncture in managing fatigue in women with breast cancer.

PURPOSE: This randomized phase III trial is studying acupuncture to see how well it works compared with self-acupuncture in managing cancer-related fatigue in women who have received chemotherapy for stage I, stage II, or stage IIIA breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Assess the efficacy of a course of acupuncture in the management of cancer-related fatigue in a homogeneous sample of women with stage I, II, or IIIA breast cancer who have completed adjuvant chemotherapy.
* Assess the efficacy of self-acupuncture in comparison to therapist-administered acupuncture in sustaining, in the longer term, any effects observed with a 6-week course of acupuncture in these patients.

OUTLINE: This is a multicenter study. Patients are stratified according to study center and fatigue score (low vs moderate vs severe). Patients are randomized at 3:1 ratio (arm I: arm II) to 1 of 2 treatment arms.

* Arm I (experimental): Patients undergo a 20-minute acupuncture session once a week for 6 weeks. Patients also receive written information about fatigue and its possible management.
* Arm II (control): Patients undergo standard care. They also receive written information about fatigue as in arm I.

After 6 weeks, patients in arm I are again randomized to 1 of 3 arms.

* Arm A: Patients receive treatment as in arm I for 4 more weeks.
* Arm B: Patients receive treatment as in arm II for 4 more weeks.
* Arm C: Patients learn to self-acupuncture and do so weekly for 4 more weeks. All patients complete questionnaires on fatigue, hospital anxiety and depression, quality of life, and use of complementary therapies at baseline and periodically during study. Patient's sociodemographic and treatment characteristic records are also reviewed.

After completion of study therapy, patients are followed up periodically for 18 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of breast cancer

  * Stage I, II, or IIIA disease
* Completed prior chemotherapy for ≥ 1 month and up to 5 years

  * No needling on the ipsilateral arm of patients who have undergone axillary dissection
  * No needling on the lymphedematous limbs
* Score of ≥ 5 on a 0-10 single-item screening fatigue scale, where 0 is no fatigue at all and 10 is extremely fatigued
* Hormone receptor status not specified

PATIENT CHARACTERISTICS:

* Life expectancy ≥ 6 months
* Menopausal status not specified
* Platelet count ≥ 50,000/mm^3
* Hemoglobin ≥ 10 g/dL
* Hematocrit ≥ 30%
* Not pregnant
* No needle phobia
* No co-morbidity with any of the following:

  * Bleeding disorder
  * Thyroid dysfunction

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No planned concurrent chemoradiotherapy
* No concurrent steroids
* No concurrent epoetin alfa or transfusion for anemia
* No other concurrent complementary therapies

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2007-10; Primary Completion 2010-10 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
General fatigue as measured by the Multidimensional Fatigue Inventory

SECONDARY OUTCOMES:
Mental fatigue as measured by the Multidimensional Fatigue Inventory
Anxiety as measured by the Hospital Anxiety and Depression Scale
Depression as measured by the Hospital Anxiety and Depression Scale
Quality of life as measured by the FACT-G and Breast Cancer module

CONTACTS AND LOCATIONS:
Overall Officials: Alex Molassiotis, MD, Principal Investigator — University of Manchester
Locations (1):
- University of Manchester, Manchester, England, United Kingdom

REFERENCES:
- [Derived] Molassiotis A, Bardy J, Finnegan-John J, Mackereth P, Ryder WD, Filshie J, Ream E, Eaton D, Richardson A. A randomized, controlled trial of acupuncture self-needling as maintenance therapy for cancer-related fatigue after therapist-delivered acupuncture. Ann Oncol. 2013 Jun;24(6):1645-52. doi: 10.1093/annonc/mdt034. Epub 2013 Feb 21. PMID 23436910
- [Derived] Molassiotis A, Bardy J, Finnegan-John J, Mackereth P, Ryder DW, Filshie J, Ream E, Richardson A. Acupuncture for cancer-related fatigue in patients with breast cancer: a pragmatic randomized controlled trial. J Clin Oncol. 2012 Dec 20;30(36):4470-6. doi: 10.1200/JCO.2012.41.6222. Epub 2012 Oct 29. PMID 23109700